CLINICAL TRIAL: NCT05886231
Title: Evaluation of Music Effects on Intraoperative and Postoperative Parameters
Brief Title: The Effects of Instrumental Music on Intraoperative Parameters and Postoperative Pain and Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023/1
Record Dates: First submitted 2023-05-13; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Music and Anesthesia
Keywords: music; anesthesia; Train of four; Bispectral index

STUDY DESIGN:
Intervention Model Description: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- music group (Group M) (Experimental): Group M patients were fitted with headphones that covered the entire ear and suppressed hearing of the sounds in the operating room. The level of the music sound was adjusted to the level where patients felt comfortable by asking them before induction.
  Mean arterial pressure (MAP) greater than 20% of the initial value for one minute or longer was first evaluated in favor of superficial anesthesia, while its continuation was considered hypertension.
  If the TOF value was higher than 70 for a long time, 0.1 mg/kg rocuronium iv was administered, and 50 µg fentanyl iv was administered in the need for opioids. In the last 20 minutes of the surgical period, 1 mg/kg tramadol and 20 mg/kg paracetamol IV were administered to all patients in accordance with conventional treatment for postoperative analgesia.
  Interventions: Other: music sound therapy

INTERVENTIONS:
Other: music sound therapy — investigate the effects of music on intraoperative hemodynamic parameters, anesthesia depth, muscle relaxant consumption, analgesic consumption and pain and side effects (nausea, vomiting, tremor) in the early postoperative period in patients undergoing thyroidectomy operation under general anesthesia.

SUMMARY:
The clinical study started after receiving ethical approval from the Clinical Research Ethics Committee of Van Yüzüncü Yıl University and obtaining patient consent. Eighty patients with an ASA (American Society of Anesthesiologists) I-II physical status at the ages of 20-60 for whom elective thyroidectomy surgery was planned were included in the study. The patients were randomly divided into two groups, music group (Group M) and control group (Group K). The intraoperative vital signs of the patients (heart rate, blood pressure and saturation), bispectral index (BIS) values, train-of-four (TOF) values, additional doses of opioid and muscle relaxant needs and complications were recorded. The 0th hour, 3rd hour and 6th hour Visual Analogue Scale (VAS) scores of the patients were measured and recorded. (The 0th hour at the end of the operation was accepted as the moment of reaching a Modified Aldrete Score of >9)

DETAILED DESCRIPTION:
This study was conducted at Yüzüncü Yıl University Dursun Odabaş Medical Center after the approval of Van Yüzüncü Yıl University Non-Interventional Clinical Research Ethics Committee and the verbal and written consent of the patients.

2.1. Population Patients with ASA I-II functional status, aged 20-60 years, who agreed to participate in the study and were scheduled for thyroidectomy under general anesthesia under elective conditions were included. Patients with emergency and bleeding, those who would undergo other surgery, those who refused to participate in the study, those with hearing problems, those who could not cooperate (due to dementia, mental retardation, etc.), those with drug or alcohol addiction, and obese patients with a BMI≥30 were excluded from the study. The patients were randomly divided into two groups as music group (Group M) and control group (Group K) by sealed tender. 40 patients in each group and a total of 80 patients were included in the study. Closed envelopes determining which group the patient would belong to were randomly selected by the patient. The patients who would participate in the study were evaluated preoperatively in the Anesthesiology and Reanimation outpatient clinic the day before and were informed about the study. Except for routine preoperative evaluation tests (hemogram, fasting blood sugar, sodium, potassium, calcium, urea, creatinine, AST (aspartate aminotransferase), ALT (alanine aminotransferase), coagulation parameters), no additional tests were requested.

The demographic data (age, weight, height, gender, body mass index (BMI)) of the patients were recorded.

2.2. Anesthesia Management Routine standard ASA monitoring electrocardiography (ECG), peripheral oxygen saturation (SpO2), heart rate (HR), non-invasive blood pressure monitoring), bispectral index monitoring (A-2000 Aspect medical systems, USA), and neuromuscular monitoring (TOF) were performed Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (map), heart rate (HR), SpO2, BIS, and TOF values were recorded. Initial values before surgery -5th-minute values were accepted and the values were recorded as of the 0th minute after the surgical incision. Measurements were taken at 5 minutes intervals in the first half hour after the start of surgery, and then at 10 minutes intervals.After the patients were placed in the appropriate position, Group M patients were fitted with headphones that covered the entire ear and suppressed hearing of the sounds in the operating room. The level of the music sound was adjusted to the level where patients felt comfortable by asking them before induction. Until the anesthetic gases ceased, relaxing instrumental classical music which is selected by us and recorded on the SD card, was played during the entire operation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II functional status,
* 20-60 years
* agreed to participate in the study
* scheduled for thyroidectomy under general anesthesia

Exclusion Criteria:

* emergence cases
* bleeding cases
* other surgeries
* refused to participate in the study,
* have hearing problems
* could not cooperate (due to dementia, mental retardation, etc.)
* drug or alcohol addiction,
* obese patients with a BMI≥30

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
heart rate | 1 day of surgery
  intraoperative vital signs of the patients (heart rate)
non invasive blood pressure | 1 day of surgery
  intraoperative vital signs of the patients ( non invasive blood pressure)
Pulse oxymeter | 1 day of surgery
  Intraoperative measurements
BIS (Bispektral index) | 15 minutes
  For monitoring being awake
level of opioid | 30 minutes
  additional opioid
muscle relaxant | 40 minutes
  additional muscle relaxant

SECONDARY OUTCOMES:
Side effects | 0., 3., 6. hours
  The patients were followed up for side effects
VAS scores | Postoperative 0th hour (0th hour was considered as the moment when Modified Aldrete Score >9), 3rd hour, and 6th- hour VAS scores of all cases were recorded.
  VAS 0-2: no pain, 3-4: dull pain, 5-6: moderate pain, 7-8: acute pain, 9-10: unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yüzüncu Yıl University Medicine School, Study Chair — Yuzuncu Yil University
Locations (2):
- Turkey (Türkiye) (2):
  - Arzu Esen Tekeli, Van
  - Van Yüzüncü Yil University, Van

IPD SHARING:
Plan to Share IPD: No
This is a retrospective study. We will share our results. W e dont plan to share participiants values